CLINICAL TRIAL: NCT04975607
Title: Live Music Therapy to Reduce Anxiety, Pain and Improve Sleep in Post-Operative Lung Transplant Patients: a Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Emily Pickett, Unit Based Educator for Clinical Care, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STU-2019-1409
Record Dates: First submitted 2021-07-01; First posted 2021-07-23 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-02

CONDITIONS: Lung Transplant; Complications
MeSH Terms: interventions — Music Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Music Therapy Group (Experimental)
  Interventions: Behavioral: Music Therapy
- Control Group (No Intervention)

INTERVENTIONS:
Behavioral: Music Therapy — The three live music therapy sessions will be provided after lung transplant. All three music therapy sessions will employ a variety of data-based interventions to address pain, anxiety, and improve relaxation. Music therapy interventions may include patient preferred live music, active music listening, singing or other active music-making, and guided breathing and relaxation.
  Arms: Music Therapy Group

SUMMARY:
The purpose of this prospective pilot study is to determine if live music therapy reduces patients' perception of pain and anxiety, reduces benzodiazepine use and pain medication use, length of stay in the ICU, and length of stay in hospital, and improves sleep in post-lung transplant patients.

The purpose and objectives of the study are the following:

* To determine if music therapist delivered patient preferred live music and therapeutic intervention will reduce participant's perceived anxiety in post-lung transplant patients.
* To determine if music therapist delivered patient preferred live music and therapeutic intervention will reduce participant's perceived pain in post-lung transplant patients.
* To determine if music therapist delivered patient preferred live music and therapeutic intervention in post-lung transplant patients will reduce participant's use of benzodiazepine medication for anxiety.
* To determine if music therapist delivered patient preferred live music and therapeutic intervention three times in post-lung transplant patients will reduce participant's use of pain medication.
* To determine if music therapist delivered patient preferred live music and therapeutic intervention in post-lung transplant patients will reduce participant's total time of intubation, length of stay in ICU, and length of stay in the hospital.
* To determine if music therapist delivered patient preferred live music and therapeutic intervention will improve the quality and length of sleep in post-lung transplant patients.

ELIGIBILITY:
Inclusion Criteria:

* All post-lung transplant patients at UTSW Clements University Hospital starting June 1, 2021

Exclusion Criteria:

* Post-lung transplant patients with chests left open directly after OR (before being taken back to the OR and having their chests closed)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2023-04-11 (Actual); Study Completion 2023-04-11 (Actual)

PRIMARY OUTCOMES:
Change in Anxiety levels | Changes from baseline to post-surgery day 6
  Comparing the scores from the Hamilton Anxiety Rating Scale (HAM-A) scale before and after music therapy. Scores range between 0-56 where <17 indicates mild severity, 18-24 mild to moderate severity and 25-30 moderate to severe.
Change in Pain levels (CPOT) | Changes from baseline to post-surgery day 6
  Comparing the scores from the Critical Care Pain Observation Tool (CPOT) scale before and after music therapy. Scores ranges between 0 (no pain) to 8 (maximum pain).
Change in Pain levels (Pain number scale) | Changes from baseline to post-surgery day 6
  Comparing the scores from the Pain number scale before and after music therapy. Scores ranges between 0 (no pain) to 10 (maximum pain).
Change in dosage of benzodiazepine medication | Changes from baseline to post-surgery day 6
  Comparing medication dosage between intervention group vs control group.
Change in dosage of pain medication | Changes from baseline to post-surgery day 6
  Comparing medication dosage between intervention group vs control group
Change in length of sleep | Changes from baseline to post-surgery day 6
  Comparing Fitbit data on length of sleep between intervention group vs control group
Change in length of stay in ICU and in hospital | Changes from baseline to post-surgery day 6
  Comparing length of stay between intervention group vs control group
Change in total time of intubation | Intubation prior to surgery until extubation (Post-surgery day 4)
  Comparing duration of intubation between intervention group vs control group

CONTACTS AND LOCATIONS:
Overall Officials: Emily Pickett, Principal Investigator — University of Texas Southwestern Medical Center; Daniel Tague, PhD, Principal Investigator — Southern Methodist University
Locations (1):
- University of Texas Southwestern Medical Center, Dallas, Texas, United States